CLINICAL TRIAL: NCT04415463
Title: EsophageAl mulTisegmented Fully covERed Self-expandable Metal Stent for Malignant Strictures: a Safety and Feasibility Study (EATERS Study)
Brief Title: Esophageal Multisegmented FCSEMS for Malignant Strictures
Acronym: EATERS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Safety concerns
Sponsor: Radboud University Medical Center (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL73180.091.20
Record Dates: First submitted 2020-05-25; First posted 2020-06-04 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Oesophageal Cancer; Esophageal Stent Stenosis
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FC-SEMS (Experimental): Placement of multisegmented fully covered self-expandable metal stent
  Interventions: Device: Multisegmented fully covered self-expandable metal stent

INTERVENTIONS:
Device: Multisegmented fully covered self-expandable metal stent — Esophageal FC-SEMS

SUMMARY:
Objective: To assess the safety and feasibility of the implementation of the esophageal multisegmented fully covered self-expandable metal stent (SEMS) for the palliation of patients with malignant dysphagia.

Study design: Prospective observational nonrandomized clinical study.

Study population: A total of 30 patients with malignant dysphagia will be included. Sample size calculation does not apply for this type of study.

Intervention: All patients will be treated with the esophageal multisegmented fully covered SEMS.

Primary end points:

* Safety: complications and adverse events during follow-up with special attention to stent migration rates;
* Efficacy: technical success of stent placement.

Secondary end points:

* Recurrent dysphagia including its cause;
* Functional outcome: Ogilvie dysphagia score and WHO performance score (measured at baseline, 2 weeks and every 4 weeks until death/stent removal, or until a maximum of 6 months follow-up);
* Tissue ingrowth or overgrowth (measured endoscopically every endoscopic evaluation during follow-up);
* Pain related to esophageal stent.

ELIGIBILITY:
Inclusion criteria:

* Patients presenting with dysphagia due to a non-operable malignant obstruction of the esophagus or esophagogastric junction including extrinsic malignant compression and recurrence in post-esophagectomy patients;
* Requiring treatment for dysphagia (Ogilvie score of 2-41);
* Life expectancy of less than 12 months.

Exclusion criteria:

* Stenosis after laryngectomy;
* Distance between the upper edge of the stent less than 2 cm from the upper esophageal sphincter;
* Esophageal fistula;
* Tumor length of more than 14 cm;
* Previous stent placement for the same condition;
* Inappropriate cultural level and understanding of the study;
* Coagulopathy;
* Patients with eosinophilic esophagitis or an esophageal motility disorder;
* Nickel titanium (Nitinol) allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | 6 months
  Adverse events during follow-up
Technical success of stent placement | 1 day
  Technical success of stent placement

SECONDARY OUTCOMES:
Recurrent dysphagia | 6 months
  Ogilvie dysphagia score
Functional outcome | 6 months
  WHO performance score
Tissue ingrowth or overgrowth | 6 months
Pain related to esophageal stent | 6 months
  Measured using the Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koggel LM, Reijm AN, Lantinga MA, de Jong DJ, Rodrigues-Pinto E, Spaander MCW, Siersema PD. Multisegmented esophageal fully covered self-expandable metal stent for palliation of malignant dysphagia: a prospective, multicenter feasibility and safety study. Gastrointest Endosc. 2024 Jun;99(6):1027-1031.e6. doi: 10.1016/j.gie.2024.01.045. Epub 2024 Feb 3. PMID 38316224